CLINICAL TRIAL: NCT01428050
Title: Prospective Randomized Controlled Trial on the Use of a Restrictive Fluid Regimen With Hypertonic Saline for Patients Undergoing Pancreaticoduodenectomy
Brief Title: The Use of a Restrictive Fluid Regimen With Hypertonic Saline for Patients Undergoing Pancreaticoduodenectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Jefferson Hypertonic
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Pancreaticoduodenectomy
Keywords: whipple; hypertonic saline; pancreaticoduodenectomy; fluid restriction; resuscitation strategy
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3% saline (Experimental): Patients will received 3% saline in conjunction with lactated ringers solution intra and post operatively for a net reduction in total fluid administration
  Interventions: Drug: 3% NaCl Solution
- Lactated Ringers (Active Comparator): 15cc/kg/hr of lactated ringers solution intraoperatively
  Interventions: Drug: Lactated Ringers Solution

INTERVENTIONS:
Drug: 3% NaCl Solution — 1cc/kg/hr of 3%NaCl + 9cc/kg/hr of lactated ringers solution
  Arms: 3% saline
Drug: Lactated Ringers Solution — 15cc/kg/hr for intraoperative fluids
  Arms: Lactated Ringers

SUMMARY:
The Whipple operation is a complex surgical procedure involving the removal of the head of the pancreas, bile duct, and a portion of the intestine (duodenum) that is performed for patients who have cancer or some other condition affecting this region of the body. The Whipple operation is associated with a significant complication rate. Previous studies have shown that in a broad range of surgical procedures, using a reduced amount of intravenous fluids along with a special type of fluid called hypertonic saline during and after the procedure can lower complication rates associated with the heart and lungs during recovery from surgery. The purpose of this study is to determine if using a reduced amount of intravenous fluids as well as hypertonic saline (a salt concentrated form of intravenous fluids) during the Whipple operation and in the immediate period after surgery can reduce complications.

ELIGIBILITY:
Inclusion Criteria:

* Physiologic suitability for major abdominal surgery
* Aged 18 years and older
* Written informed consent
* Ability to understand and comply with study guidelines
* Ability to obtain a central venous line

Exclusion Criteria:

* Metabolic acidosis
* Active Sepsis or Bacteremia
* Chronic renal insufficiency
* Hyponatremia (serum sodium <130)
* Hypernatremia (serum sodium >150)
* Pregnancy
* Sickle cell anemia
* Pediatric patients
* BMI>40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2011-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Anastomotic Leak | 30 days
  Leak or defect of gastrointestinal anastomosis including but not limited to pancreaticojejunostomy
Delayed Gastric Emptying | 30 days
  Rate of delayed gastric emptying post procedure, prolonged initiation of enteral feeding
Myocardial Infarction | 30 days
Pneumonia | 30 days
Wound Infection | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Harish Lavu, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Lavu H, Sell NM, Carter TI, Winter JM, Maguire DP, Gratch DM, Berman RA, Feil MG, Grunwald Z, Leiby BE, Pequignot EC, Rosato EL, Yeo CJ. The HYSLAR trial: a prospective randomized controlled trial of the use of a restrictive fluid regimen with 3% hypertonic saline versus lactated Ringers in patients undergoing pancreaticoduodenectomy. Ann Surg. 2014 Sep;260(3):445-53; discussion 453-5. doi: 10.1097/SLA.0000000000000872. PMID 25115420